CLINICAL TRIAL: NCT03959371
Title: Observational, Retrospective and Prospective Study on the Use of Ruxolitinib in Myelofibrosis Patients in Lombardy, Italy
Brief Title: Ruxolitinib in Myelofibrosis Patients in Lombardy, Italy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Margherita Maffioli (Other)
Responsible Party: Sponsor-Investigator, Margherita Maffioli, Principal Investigator, Ospedale di Circolo - Fondazione Macchi
Organization: Ospedale di Circolo - Fondazione Macchi (Other)
Other Study IDs: RUXOREL-MF
Record Dates: First submitted 2019-04-07; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Ruxolitinib; Real world data
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ruxolitinib — Observational study including patients with myelofibrosis being treated with ruxolitinib in a "real world" setting. Patients are treated according to current indications.

SUMMARY:
The RUXOREL-MF observational study includes patients with primary and post-essential thrombocythemia/post-polycythemia vera myelofibrosis (MF) being treated with the oral JAK1-/JAK2-inhibitor ruxolitinib in a "real world" setting. Patients are treated according to current indications in Italy (i.e., primary and secondary MF patients with intermediate-1, intermediate-2, and high risk IPSS (International Prognostic Scoring System) scores and symptomatic splenomegaly and/or systemic symptoms). Patients are treated at facilities pertaining to the regional Hematology Network of Lombardy (Rete Ematologica Lombarda) in Italy. Efficacy data, data related to infectious and vascular events, data related to second primary malignancies, data regarding disease progression/transformation, and molecular information in relationship to ruxolitinib treatment will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of primary myelofibrosis diagnosis according to the WHO 2016 classification or post-essential thrombocythemia/post-polycythemia vera myelofibrosis according to the IWG-MRT 2008 classification
* Patients with an intermediate-1, intermediate-2, or high risk score according to the IPSS (International Prognostic Scoring System)
* Patients treated with ruxolitinib in accordance with current indications in Italy
* Patients eligible or ineligible to hematopoietic stem cell transplant or who have already undergone a hematopoietic stem cell transplant

Exclusion Criteria:

* Diagnoses other than primary myelofibrosis or post-essential thrombocythemia/post-polycythemia vera myelofibrosis
* Patients treated with ruxolitinib having a platelet count at treatment initiation <50 x10^9/L
* Patients treated with ruxolitinib for conditions other than primary myelofibrosis or post-essential thrombocythemia/post-polycythemia vera myelofibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary myelofibrosis diagnosis according to the WHO (World Health Organization) 2016 classification or post-essential thrombocythemia/post-polycythemia vera myelofibrosis diagnosis according to the IWG-MRT (International Working Group for Myelofibrosis Research and Treatment) 2008 classification, with an intermediate-1, intermediate-2, or high risk score according to the IPSS (International Prognostic Scoring System), treated with ruxolitinib in accordance with current indications in Italy and pertaining to centers of the regional Hematology Network of Lombardy (Rete Ematologica Lombarda), Italy.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of infectious events after ruxolitinib exposure in myelofibrosis patients | Through study completion, an average of 1 year
Rate of vascular events after ruxolitinib exposure in myelofibrosis patients | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Spleen response rate | At 3 and 6 months from ruxolitinib start
Rate of primary secondary malignancies | Through study completion, an average of 1 year
Acute myeloid leukemia transformation rate | Through study completion, an average of 1 year
Rate of infectious events according to driver mutational status (i.e., mutations of JAK2, CALR, or MPL) | Through study completion, an average of 1 year
  Association of rate of infectious events with driver mutational status
Rate of vascular events according to driver mutational status (i.e., mutations of JAK2, CALR, or MPL) | Through study completion, an average of 1 year
  Association of rate of vascular events with driver mutational status
Spleen response rate according to driver mutational status (i.e., mutations of JAK2, CALR, or MPL) | Through study completion, an average of 1 year
  Association of spleen response rate with driver mutational status
Rate of primary secondary malignancies according to driver mutational status (i.e., mutations of JAK2, CALR, or MPL) | Through study completion, an average of 1 year
  Association of rate of primary secondary malignancies with driver mutational status
Acute myeloid leukemia transformation rate according to driver mutational status (i.e., mutations of JAK2, CALR, or MPL) | Through study completion, an average of 1 year
  Association of acute myeloid leukemia transformation rate with driver mutational status
Rate of infectious events according to the presence of additional mutations | Through study completion, an average of 1 year
  Association of rate of infectious events with the presence of additional mutations
Rate of vascular events according to the presence of additional mutations | Through study completion, an average of 1 year
  Association of rate of vascular events with the presence of additional mutations
Spleen response rate according to the presence of additional mutations | Through study completion, an average of 1 year
  Association of spleen response rate with the presence of additional mutations
Rate of primary secondary malignancies according to the presence of additional mutations | Through study completion, an average of 1 year
  Association of rate of primary secondary malignancies with the presence of additional mutations
Acute myeloid leukemia transformation rate according to the presence of additional mutations | Through study completion, an average of 1 year
  Association of acute myeloid leukemia transformation rate with the presence of additional mutations
Evaluation of overall survival after ruxolitinib start and, if applicable, discontinuation | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Passamonti, MD, Principal Investigator — Ospedale di Circolo ASST Sette Laghi, Università dell'Insubria, Varese, Italy
Locations (12):
- Italy (12):
  - ASST Papa Giovanni XXIII, Bergamo
  - U.O. Ematologia, ASST Spedali Civili, Brescia
  - U.S.D. Trapianti di Midollo Osseo, ASST Spedali Civili, Brescia
  - U.O.C. di Ematologia Clinica, ASST Lecco, Lecco
  - U.O. Ematologia, ASST Fatebenefratelli-Sacco, Milan
  - U.O. Ematologia, Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - U.O. Ematologia, Grande Ospedale Metropolitano Niguarda, Milan
  - U.O. Ematologia, Humanicas Cancer Center, Milan
  - U.O. Ematologia, Ospedale San Raffaele, Milan
  - U.O. Oncoematologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Clinica Ematologica, Ospedale San Gerardo, Monza
  - Ospedale di Circolo, ASST Sette Laghi, Varese

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Barosi G, Mesa RA, Thiele J, Cervantes F, Campbell PJ, Verstovsek S, Dupriez B, Levine RL, Passamonti F, Gotlib J, Reilly JT, Vannucchi AM, Hanson CA, Solberg LA, Orazi A, Tefferi A; International Working Group for Myelofibrosis Research and Treatment (IWG-MRT). Proposed criteria for the diagnosis of post-polycythemia vera and post-essential thrombocythemia myelofibrosis: a consensus statement from the International Working Group for Myelofibrosis Research and Treatment. Leukemia. 2008 Feb;22(2):437-8. doi: 10.1038/sj.leu.2404914. Epub 2007 Aug 30. No abstract available. PMID 17728787
- [Background] Caramazza D, Begna KH, Gangat N, Vaidya R, Siragusa S, Van Dyke DL, Hanson C, Pardanani A, Tefferi A. Refined cytogenetic-risk categorization for overall and leukemia-free survival in primary myelofibrosis: a single center study of 433 patients. Leukemia. 2011 Jan;25(1):82-8. doi: 10.1038/leu.2010.234. Epub 2010 Oct 14. PMID 20944670
- [Background] Cervantes F, Dupriez B, Pereira A, Passamonti F, Reilly JT, Morra E, Vannucchi AM, Mesa RA, Demory JL, Barosi G, Rumi E, Tefferi A. New prognostic scoring system for primary myelofibrosis based on a study of the International Working Group for Myelofibrosis Research and Treatment. Blood. 2009 Mar 26;113(13):2895-901. doi: 10.1182/blood-2008-07-170449. Epub 2008 Nov 6. PMID 18988864
- [Background] Cervantes F, Vannucchi AM, Kiladjian JJ, Al-Ali HK, Sirulnik A, Stalbovskaya V, McQuitty M, Hunter DS, Levy RS, Passamonti F, Barbui T, Barosi G, Harrison CN, Knoops L, Gisslinger H; COMFORT-II investigators. Three-year efficacy, safety, and survival findings from COMFORT-II, a phase 3 study comparing ruxolitinib with best available therapy for myelofibrosis. Blood. 2013 Dec 12;122(25):4047-53. doi: 10.1182/blood-2013-02-485888. Epub 2013 Oct 30. PMID 24174625
- [Background] Gangat N, Caramazza D, Vaidya R, George G, Begna K, Schwager S, Van Dyke D, Hanson C, Wu W, Pardanani A, Cervantes F, Passamonti F, Tefferi A. DIPSS plus: a refined Dynamic International Prognostic Scoring System for primary myelofibrosis that incorporates prognostic information from karyotype, platelet count, and transfusion status. J Clin Oncol. 2011 Feb 1;29(4):392-7. doi: 10.1200/JCO.2010.32.2446. Epub 2010 Dec 13. PMID 21149668
- [Background] Guglielmelli P, Biamonte F, Rotunno G, Artusi V, Artuso L, Bernardis I, Tenedini E, Pieri L, Paoli C, Mannarelli C, Fjerza R, Rumi E, Stalbovskaya V, Squires M, Cazzola M, Manfredini R, Harrison C, Tagliafico E, Vannucchi AM; COMFORT-II Investigators; Associazione Italiana per la Ricerca sul Cancro Gruppo Italiano Malattie Mieloproliferative (AGIMM) Investigators. Impact of mutational status on outcomes in myelofibrosis patients treated with ruxolitinib in the COMFORT-II study. Blood. 2014 Apr 3;123(14):2157-60. doi: 10.1182/blood-2013-11-536557. Epub 2014 Jan 23. PMID 24458439
- [Background] Guglielmelli P, Lasho TL, Rotunno G, Mudireddy M, Mannarelli C, Nicolosi M, Pacilli A, Pardanani A, Rumi E, Rosti V, Hanson CA, Mannelli F, Ketterling RP, Gangat N, Rambaldi A, Passamonti F, Barosi G, Barbui T, Cazzola M, Vannucchi AM, Tefferi A. MIPSS70: Mutation-Enhanced International Prognostic Score System for Transplantation-Age Patients With Primary Myelofibrosis. J Clin Oncol. 2018 Feb 1;36(4):310-318. doi: 10.1200/JCO.2017.76.4886. Epub 2017 Dec 9. PMID 29226763
- [Background] Harrison C, Kiladjian JJ, Al-Ali HK, Gisslinger H, Waltzman R, Stalbovskaya V, McQuitty M, Hunter DS, Levy R, Knoops L, Cervantes F, Vannucchi AM, Barbui T, Barosi G. JAK inhibition with ruxolitinib versus best available therapy for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):787-98. doi: 10.1056/NEJMoa1110556. PMID 22375970
- [Background] Harrison CN, Vannucchi AM, Kiladjian JJ, Al-Ali HK, Gisslinger H, Knoops L, Cervantes F, Jones MM, Sun K, McQuitty M, Stalbovskaya V, Gopalakrishna P, Barbui T. Long-term findings from COMFORT-II, a phase 3 study of ruxolitinib vs best available therapy for myelofibrosis. Leukemia. 2016 Aug;30(8):1701-7. doi: 10.1038/leu.2016.148. Epub 2016 May 23. PMID 27211272
- [Background] Heine A, Brossart P, Wolf D. Ruxolitinib is a potent immunosuppressive compound: is it time for anti-infective prophylaxis? Blood. 2013 Nov 28;122(23):3843-4. doi: 10.1182/blood-2013-10-531103. No abstract available. PMID 24288410
- [Background] Kroger NM, Deeg JH, Olavarria E, Niederwieser D, Bacigalupo A, Barbui T, Rambaldi A, Mesa R, Tefferi A, Griesshammer M, Gupta V, Harrison C, Alchalby H, Vannucchi AM, Cervantes F, Robin M, Ditschkowski M, Fauble V, McLornan D, Ballen K, Popat UR, Passamonti F, Rondelli D, Barosi G. Indication and management of allogeneic stem cell transplantation in primary myelofibrosis: a consensus process by an EBMT/ELN international working group. Leukemia. 2015 Nov;29(11):2126-33. doi: 10.1038/leu.2015.233. Epub 2015 Aug 21. PMID 26293647
- [Background] Newberry KJ, Patel K, Masarova L, Luthra R, Manshouri T, Jabbour E, Bose P, Daver N, Cortes J, Kantarjian H, Verstovsek S. Clonal evolution and outcomes in myelofibrosis after ruxolitinib discontinuation. Blood. 2017 Aug 31;130(9):1125-1131. doi: 10.1182/blood-2017-05-783225. Epub 2017 Jul 3. PMID 28674026
- [Background] Passamonti F, Maffioli M. Update from the latest WHO classification of MPNs: a user's manual. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):534-542. doi: 10.1182/asheducation-2016.1.534. PMID 27913526
- [Background] Passamonti F, Cervantes F, Vannucchi AM, Morra E, Rumi E, Pereira A, Guglielmelli P, Pungolino E, Caramella M, Maffioli M, Pascutto C, Lazzarino M, Cazzola M, Tefferi A. A dynamic prognostic model to predict survival in primary myelofibrosis: a study by the IWG-MRT (International Working Group for Myeloproliferative Neoplasms Research and Treatment). Blood. 2010 Mar 4;115(9):1703-8. doi: 10.1182/blood-2009-09-245837. Epub 2009 Dec 14. PMID 20008785
- [Background] Passamonti F, Mora B, Giorgino T, Guglielmelli P, Cazzola M, Maffioli M, Rambaldi A, Caramella M, Komrokji R, Gotlib J, Kiladjian JJ, Cervantes F, Devos T, Palandri F, De Stefano V, Ruggeri M, Silver R, Benevolo G, Albano F, Caramazza D, Rumi E, Merli M, Pietra D, Casalone R, Barbui T, Pieri L, Vannucchi AM. Driver mutations' effect in secondary myelofibrosis: an international multicenter study based on 781 patients. Leukemia. 2017 Apr;31(4):970-973. doi: 10.1038/leu.2016.351. Epub 2016 Nov 25. No abstract available. PMID 27885272
- [Background] Passamonti F, Giorgino T, Mora B, Guglielmelli P, Rumi E, Maffioli M, Rambaldi A, Caramella M, Komrokji R, Gotlib J, Kiladjian JJ, Cervantes F, Devos T, Palandri F, De Stefano V, Ruggeri M, Silver RT, Benevolo G, Albano F, Caramazza D, Merli M, Pietra D, Casalone R, Rotunno G, Barbui T, Cazzola M, Vannucchi AM. A clinical-molecular prognostic model to predict survival in patients with post polycythemia vera and post essential thrombocythemia myelofibrosis. Leukemia. 2017 Dec;31(12):2726-2731. doi: 10.1038/leu.2017.169. Epub 2017 May 31. PMID 28561069
- [Background] Rotunno G, Pacilli A, Artusi V, Rumi E, Maffioli M, Delaini F, Brogi G, Fanelli T, Pancrazzi A, Pietra D, Bernardis I, Belotti C, Pieri L, Sant'Antonio E, Salmoiraghi S, Cilloni D, Rambaldi A, Passamonti F, Barbui T, Manfredini R, Cazzola M, Tagliafico E, Vannucchi AM, Guglielmelli P. Epidemiology and clinical relevance of mutations in postpolycythemia vera and postessential thrombocythemia myelofibrosis: A study on 359 patients of the AGIMM group. Am J Hematol. 2016 Jul;91(7):681-6. doi: 10.1002/ajh.24377. Epub 2016 May 11. PMID 27037840
- [Background] Rumi E, Pietra D, Pascutto C, Guglielmelli P, Martinez-Trillos A, Casetti I, Colomer D, Pieri L, Pratcorona M, Rotunno G, Sant'Antonio E, Bellini M, Cavalloni C, Mannarelli C, Milanesi C, Boveri E, Ferretti V, Astori C, Rosti V, Cervantes F, Barosi G, Vannucchi AM, Cazzola M; Associazione Italiana per la Ricerca sul Cancro Gruppo Italiano Malattie Mieloproliferative Investigators. Clinical effect of driver mutations of JAK2, CALR, or MPL in primary myelofibrosis. Blood. 2014 Aug 14;124(7):1062-9. doi: 10.1182/blood-2014-05-578435. Epub 2014 Jul 1. PMID 24986690
- [Background] Spiegel JY, McNamara C, Kennedy JA, Panzarella T, Arruda A, Stockley T, Sukhai M, Thomas M, Bartoszko J, Ho J, Siddiq N, Maze D, Schimmer A, Schuh A, Sibai H, Yee K, Claudio J, Devlin R, Minden MD, Kamel-Reid S, Gupta V. Impact of genomic alterations on outcomes in myelofibrosis patients undergoing JAK1/2 inhibitor therapy. Blood Adv. 2017 Sep 8;1(20):1729-1738. doi: 10.1182/bloodadvances.2017009530. eCollection 2017 Sep 12. PMID 29296819
- [Background] Thiele J, Kvasnicka HM, Facchetti F, Franco V, van der Walt J, Orazi A. European consensus on grading bone marrow fibrosis and assessment of cellularity. Haematologica. 2005 Aug;90(8):1128-32. PMID 16079113
- [Background] Vannucchi AM, Kantarjian HM, Kiladjian JJ, Gotlib J, Cervantes F, Mesa RA, Sarlis NJ, Peng W, Sandor V, Gopalakrishna P, Hmissi A, Stalbovskaya V, Gupta V, Harrison C, Verstovsek S; COMFORT Investigators. A pooled analysis of overall survival in COMFORT-I and COMFORT-II, 2 randomized phase III trials of ruxolitinib for the treatment of myelofibrosis. Haematologica. 2015 Sep;100(9):1139-45. doi: 10.3324/haematol.2014.119545. Epub 2015 Jun 11. PMID 26069290
- [Background] Vannucchi AM, Lasho TL, Guglielmelli P, Biamonte F, Pardanani A, Pereira A, Finke C, Score J, Gangat N, Mannarelli C, Ketterling RP, Rotunno G, Knudson RA, Susini MC, Laborde RR, Spolverini A, Pancrazzi A, Pieri L, Manfredini R, Tagliafico E, Zini R, Jones A, Zoi K, Reiter A, Duncombe A, Pietra D, Rumi E, Cervantes F, Barosi G, Cazzola M, Cross NC, Tefferi A. Mutations and prognosis in primary myelofibrosis. Leukemia. 2013 Sep;27(9):1861-9. doi: 10.1038/leu.2013.119. Epub 2013 Apr 26. PMID 23619563
- [Background] Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, Catalano JV, Deininger M, Miller C, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner E, Lyons RM, Paquette R, Raza A, Vaddi K, Erickson-Viitanen S, Koumenis IL, Sun W, Sandor V, Kantarjian HM. A double-blind, placebo-controlled trial of ruxolitinib for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):799-807. doi: 10.1056/NEJMoa1110557. PMID 22375971